CLINICAL TRIAL: NCT02343198
Title: The Use of NMES as a Home-based Therapy Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Galway Clinic (Network); Irish Research Council (Other)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HB_NMES_PC
Record Dates: First submitted 2015-01-12; First posted 2015-01-21 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation (Experimental): Custom-built research muscle stimulator. Muscle stimulator is set to provide a comfortable stimulation when applied to the soleus muscle using two 5x5cm electrodes.
  Interventions: Device: Custom-built research muscle stimulator
- Placebo-control (Placebo Comparator): Custom-built research muscle stimulator. Muscle stimulator is set to provide sensory stimulation but will not cause an active muscle contraction. Stimulation is also delivered to the soleus muscle through two 5x5cm electrodes.
  Interventions: Device: Custom-built research muscle stimulator

INTERVENTIONS:
Device: Custom-built research muscle stimulator — Muscle stimulator

SUMMARY:
The use of neuromuscular electrical stimulation (NMES) as a home-based therapy following total knee arthroplasty. Measures of interest: lower limb venous hemodynamics, joint range of motion, lower limb swelling, walking speed, quality of life, activities of daily living, device usability, device compliance, activity levels, and pain (VAS).

DETAILED DESCRIPTION:
The use of neuromuscular electrical stimulation (NMES) as a home-based therapy following total knee arthroplasty. All participants receive and use a research stimulator for approximately 5 weeks following total knee arthroplasty. Participants randomised to either a stimulation group or placebo-controlled group. Stimulation of the soleus muscle to investigate the effects on lower limb venous hemodynamics, joint range of motion, lower limb swelling, walking speed, quality of life, activities of daily living, device usability, device compliance, activity levels, and pain (VAS) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing knee arthroplasty in the Galway Clinic with an ability to understand the nature of the study
* Ability to give informed consent
* Not excluded based on exclusion criteria

Exclusion Criteria:

* history of symptomatic heart disease or severe arterial disease
* pregnancy
* presence of a pacemaker
* history of neurological disorder
* presence of cognitive difficulties which may prevent the patient or his/her carer from using the stimulator properly

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Lower limb venous hemodynamics using Doppler ultrasound | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  Venous hemodynamics using Doppler ultrasound

SECONDARY OUTCOMES:
Joint range of motion Knee and ankle range of motion using a goniometer | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  Knee and ankle range of motion using a goniometer
Lower limb swelling Circumference measures and volume calculations | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  Circumference measures and volume calculations
Pain (associated with stimulation) on a visual analogue scale | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  Visual analogue scale
Activity levels ActivPAL activity monitor | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  ActivPAL activity monitor
Activities of daily living Lawton, Katz, Barthel scales | One week (on average) pre-operation, 3 weeks post-operation and 6 weeks post-operation
  Lawton, Katz, Barthel scales
Quality of life QoL scales- Knee injury and Osteoarthritis Outcome Score (KOOS) | One week (on average) pre-operation, 3 weeks post-operation and 6 weeks post-operation
  QoL scales- Knee injury and Osteoarthritis Outcome Score (KOOS)
Compliance with use of the custom-built research muscle stimulator | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  Compliance with the use of the research stimulator, i.e. adherence to the stimulation protocol for both the number of sessions and the duration of stimulation for each session over the 5 weeks the stimulator is used for
Device usability System Usability Scale (SUS), Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) scales | 6 weeks post-operation
  System Usability Scale (SUS), Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) scales
Walking speed 10 metre walk test | Participants will be followed from baseline (on average one week pre-operation) up to 6 weeks post-operation
  10 metre walk test

CONTACTS AND LOCATIONS:
Overall Officials: Sandra O'Connell, B.Sc, Principal Investigator — NUI Galway, Ireland
Locations (1):
- Galway Clinic, Galway, Ireland